CLINICAL TRIAL: NCT01063959
Title: Advantages of Sleeve Gastrectomy Over Gastric Bypass for Private Pay Patients Seeking Obesity Surgery
Brief Title: Sleeve Gastrectomy Versus Gastric Bypass for Private Pay Patients Seeking Obesity Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No Enrollment
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Principal Investigator, Frank Greenway, Principal INvestigator, Pennington Biomedical Research Center
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: PBRC 294EX; FWA 00006218 (Other: Ethicon Endosurgery)
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Morbid Obesity
Keywords: Laparoscopic Sleeve Gastrectomy; Laparoscopic Gastric Bypass
MeSH Terms: conditions — Obesity, Morbid | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Safety (Other): Chart review will evaluate the safety of the two procedures, incidence of complications operatively, hospital stay, and 6-week post-operative periods.
  Interventions: Procedure: Laparoscopic Sleeve Gastrectomy; Procedure: Laparoscopic Gastric Bypass
- Weight Loss (Experimental): Chart review will evaluate weight loss in subjects during the operative, 6-week post-operative, and follow-up of at least 18 months.
  Interventions: Procedure: Laparoscopic Sleeve Gastrectomy; Procedure: Laparoscopic Gastric Bypass
- Insurance versus Private Pay (Other): An insurance company issues an insurance policy to cover specific complications from the gastric bypass or the sleeve gastrectomy surgery which allows the surgeon to offer a fixed price to the patient. Comparison of surgical complications in subjects paying by insurance versus paying personally for the gastric bypass operation.
  Interventions: Procedure: Laparoscopic Sleeve Gastrectomy; Procedure: Laparoscopic Gastric Bypass

INTERVENTIONS:
Procedure: Laparoscopic Sleeve Gastrectomy — Sleeve Gastrectomy was originally reported as the first step in an alternative two-staged procedure for the super obese patient to decrease morbidity, predominantly private pay.
  Other Names: Lap Surgery
Procedure: Laparoscopic Gastric Bypass — Presently, the laparoscopically performed gastric bypass accounts for 80% of obesity surgery in the United States, predominantly covered by insurance.
  Other Names: Gastric Bypass

SUMMARY:
The purpose of this study is to determine laparoscopic sleeve gastrectomy is a safer surgery than the gastric bypass, gives similar weight losses and that the safety of gastric in private pay patients versus insurance patients will be similar. This is a retrospective chart review of intervention charts.

DETAILED DESCRIPTION:
This study is a retrospective chart review of 800 intervention charts each for consecutive laparoscopic sleeve gastrectomies compared to consecutive laparoscopic gastric bypasses performed by two surgeons in a Louisiana private practice. This retrospective chart review will evaluate the safety of the two procedures during the operative and 6-week post-operative periods, compare the insurance patients to the private pay patients having the gastric bypass, and comparative weight loss in subjects with a follow-up of at least 18 months. This offers the unique opportunity to compare any differences in surgical complications in subjects paying by insurance versus those paying personally for the gastric bypass operation.

ELIGIBILITY:
Inclusion Criteria:

* The last 800 consecutive patients in the surgical practice of Drake Bellanger and Andrew Hargroder who had a laparoscopic sleeve gastrectomy.
* The last 800 consecutive patients in the surgical practice of Drake Bellanger and Andrew Hargroder who had a laparoscopic gastric bypass.

Exclusion Criteria:

* Subjects having any other obesity surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Comparison of the incidence of weight loss and complications operatively and in the first 6 weeks post-operatively after gastric bypass compared to sleeve gastrectomy. | 18 Months

SECONDARY OUTCOMES:
Comparison of the incidence of complications in gastric bypass patients covered by insurance vs. private pay patients during surgery, in the hospital and during the first 6 weeks post-operatively. | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Drake Bellanger, MD, Principal Investigator — Pennington Biomedial Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States